CLINICAL TRIAL: NCT03907423
Title: Effects of Rosuvastatin on Markers of Atherosclerosis in Diabetic Patients Treated With Glimepiride/Metformin Combination
Brief Title: Rosuvastatin on Diabetic Patients Treated With Glimepiride/Metformin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehab Werida (Other)
Responsible Party: Sponsor-Investigator, Rehab Werida, Principal Investigator, Damanhour University
Organization: Damanhour University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rosuvastatin on diabetics
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: T2DM.
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Metformin

STUDY DESIGN:
Intervention Model Description: Subjects will be divided into two group (one arm is DM-type 2 patients who will receive rosuvastatin -metformin-glimepiride combination (40 patients) and another arm is DM-type 2 patient who will receive glimepiride-metformin combination (30 patients).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin (Experimental): DM-type 2 patients who will receive rosuvastatin -metformin-glimepiride combination (40 patients)
  Interventions: Drug: Rosuvastatin10 mg tablet
- Placebo Group (Placebo Comparator): DM-type 2 patient who will receive glimepiride-metformin combination (30 patients).
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Rosuvastatin10 mg tablet — Diabetic patients treated with Rosuvastatin 10mg/day plus Glimepiride 1-8mg/day and Metformin 500-2550 mg/day oral
  Other Names: Glimepiride 1-8mg/day and Metformin 500-2550 mg/day oral
  Arms: Rosuvastatin
Drug: Placebo Oral Tablet — Diabetic patients treated with Glimepiride 1-8mg/day and Metformin 500-2550 mg/day oral
  Other Names: Glimepiride 1-8mg/day and Metformin 500-2550 mg/day oral
  Arms: Placebo Group

SUMMARY:
study effects of rosuvastatin on markers of atherosclerosis, thrombosis, in diabetic patients treated with glimepiride/metformin without coronary artery disease.

This effect will be investigated especially on sortilin ,fetuin-A

DETAILED DESCRIPTION:
A randomized controlled trial on 70 patients with DM type 2 will be recruited from Damanhour national medical institute.

* Subjects will be divided into two group (one arm is DM-type 2 patients who will receive rosuvastatin -metformin-glimepiride combination (40 patients) and another arm is DM-type 2 patient who will receive glimepiride-metformin combination (30 patients).
* Determination of serum levels of fetuin A and Sortilin
* Blood samples will be collected after 3-month after active treatment.
* Outcomes measurement : Sortilin ,fetuinA, Atherogenic index (AI) and coronary risk index (CRI) .

Methodology

* Sortilin, fetuinA will be determined by ELISA.
* Lipid profile.
* FBG and Hb A1C will be measured.
* Atherogenic index (AI = LDL-C/HDL-C) and CRI (CRI = TC/HDL-C) will be calculated for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus on oral therapy.
* Age 21-65 years
* Life expectancy >1 year.

Exclusion Criteria:

* Documented CVD
* Planned surgical intervention.
* Hypersensitivity to either of the study drug components.
* Type I diabetes.
* Current Insulin treatment.
* Hepatic impairment known hepatic failure.
* Inability to comply with study protocol.
* Active malignancy.
* Chronic inflammation (i.e. inflammatory bowel disease, lupus, inflammatory arthritis, rheumatoid arthritis) or chronic infection (i.e. chronic diabetic foot infection).
* Pregnancy, lactation or child-bearing potential.
* Chronic renal disease

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
serum levels of fetuin A | three months
  Fetuin-A has a diagnostic potential as a biomarker for liver dysfunction, cardiovascular diseases and disorders associated with metabolic syndrome.
serum levels of Sortilin | three months
  Sortilin is involved in lipid metabolism, promotes the development of atherosclerosis, and possibly becomes a potential therapeutic target for atherosclerosis treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass.Prof., Principal Investigator — Damanhour University
Locations (1):
- Damanhour Medical National Institute, Damanhūr, N/A = Not Appُlicable, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh TJ, Ahn CH, Kim BR, Kim KM, Moon JH, Lim S, Park KS, Lim C, Jang H, Choi SH. Circulating sortilin level as a potential biomarker for coronary atherosclerosis and diabetes mellitus. Cardiovasc Diabetol. 2017 Jul 20;16(1):92. doi: 10.1186/s12933-017-0568-9. PMID 28728579
- [Background] Dabrowska AM, Tarach JS, Wojtysiak-Duma B, Duma D. Fetuin-A (AHSG) and its usefulness in clinical practice. Review of the literature. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2015 Sep;159(3):352-9. doi: 10.5507/bp.2015.018. Epub 2015 Apr 24. PMID 25916279